CLINICAL TRIAL: NCT01607177
Title: Text Messaging to Improve Adherence to Prehabilitation in Patients Undergoing Bariatric Surgery: a Randomised Controlled Trial
Brief Title: Do Text Message Reminders Increase Preoperative Exercise in Obesity Surgery Candidates?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, SACS, Professor Andrew G. Hill, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bariatric Prehabilitation
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Perioperative Care; Bariatric Surgery; Obesity
MeSH Terms: conditions — Obesity

ARMS (2):
- Text message group (Experimental): Patients randomised to this group will receive daily text message reminders used to motivate them to exercise in the preoperative period. They will also receive an exercise information sheet to complement the text messages.
  Interventions: Behavioral: Daily text message reminders
- No text message group (No Intervention): Patients randomised to this group will receive standardised exercise advice but will not receive the text message reminders or the exercise information sheet.

INTERVENTIONS:
Behavioral: Daily text message reminders — Daily text message reminders to motivate patients to exercise in conjunction with an exercise information sheet.
  Arms: Text message group

SUMMARY:
Preoperative exercise has been shown to improve physiological and functional capacity in patients undergoing abdominal surgery to prepare them for the stress of surgery. Patients undergoing bariatric surgery are advised to partake in regular preoperative exercise. In the setting of bariatric surgery, as well as preparing patients for the stress of surgery, it is also thought to increase the likelihood that they will exercise postoperatively. However, compliance to this advice is extremely low. Text-message interventions have been shown to improve compliance to other lifestyle interventions. The investigators will compare the rate of compliance to preoperative exercise prior to bariatric surgery in patients who receive a daily text message to those who do not. The investigators will also compare weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients having laparoscopic sleeve gastrectomy at Manukau Surgery Centre
* Operation used primarily for the treatment of morbid obesity

Exclusion Criteria:

* Operation not performed at Manukau Surgery Centre
* Patient does not have a mobile phone which can receive text messages

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients partaking in the minimum recommended amount of weekly physical activity | 6 weeks post recruitment
  >450 METmins per week of physical activity as measured by the internationally and locally validated IPAQ questionnaire.

SECONDARY OUTCOMES:
Postoperative Physical Activity | 6 weeks postoperatively
  Quantity of physical acitivty will be measured as METmins per week as measured by the IPAQ questionnaire
Functional capacity | Baseline and 6 weeks post recuitment (preoperatively)
  Measured using the 6 minute walk test
Length of Hospital Stay | As assessed at day of discharge
  Total number of days spent in hospital following their operation
Short term weight loss | Out to 6 months postoperatively
  Postoperative weight loss as measured by percentage of excess weight loss
Perioperative complications | Out to 30 days postoperatively
  Prospectively recorded postoperative complications graded according the Clavien-Dindo classification system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB, MD, EdD, FRACS, FACS, Principal Investigator — South Auckland Clinical School, University of Auckland
Locations (1):
- Manukau Surgery Centre, Auckland, Manukau City, New Zealand